CLINICAL TRIAL: NCT03364933
Title: Primary Intensivists and Primary Nurses to Decrease Pediatric ICU Length of Stay
Acronym: PIPRNs
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Responsible Party: Principal Investigator, Jeffrey D. Edwards, Assistant Professor of Pediatrics, Columbia University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: AAAR5445
Record Dates: First submitted 2017-11-28; First posted 2017-12-07 (Actual); Last update posted 2020-07-27 (Actual); Status verified 2020-07

CONDITIONS: ICU Length of Stay
Keywords: Child; Critical Illness; Length of Stay; Satisfaction
MeSH Terms: conditions — Critical Illness; Personal Satisfaction | interventions — Nurses

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Primary intensivist and nurses (Experimental): Patients randomized to the experimental arm will have a primary intensivist and a team of primary nurses assigned to them.
  Interventions: Behavioral: Primary intensivist and nurses
- Control (No Intervention): Patients who are randomized to the control group will receive usual care and not be assigned a primary intensivist or nurses.

INTERVENTIONS:
Behavioral: Primary intensivist and nurses — Primary intensivist will have no active role in the daily management of patients. The primary intensivist should facilitate decision-making, be a liaison between the patient/family and PICU team, and be a resource of information for all. Responsibilities of primary intensivist:
  * Weekly check-in with and availability to patient/family
  * Attendance at family meetings
  * Availability to PICU team
  Primary nurses will be a team of up to 7 ICU nurses who will provide as much of the bedside care as possible. Responsibilities of primary nurses:
  * Maintain a primary nurse binder (paper format) for on-going communication about the patient among the team members; it will be their discretion what is information is communicated.
  * The Primary Nurse or delegate will be involved in all team/family meetings and will be expected/given an opportunity to speak during these meetings.
  Arms: Primary intensivist and nurses

SUMMARY:
This is a randomized control trial of PICU patients admitted for 7 days and expected to remain for at least another 3 days and who have a complex chronic condition. Patients will be randomized to usual care or usual care plus a primary intensivist and group of primary nurses (to facilitate passing of important patient information and informed, expedited decision-making). The primary research question is whether having a primary intensivist and nurses decreases PICU length of stay.

DETAILED DESCRIPTION:
Long-stay intensive care unit (ICU) patients, or children who require prolonged hospitalization in the pediatric ICU (PICU), represent a minority of PICU patients but have a disproportionate impact on hospital resources and unfavorable outcomes, including morbidity, mortality, and repeated critical illness. These patients and their families have multifaceted needs (eg, tailored communication) that pose unique challenges to PICU providers and the parent-provider relationship. These experiences and needs are compounded and complicated by the transitory care that is typically provided by PICU. This transitory care may contribute to 1) patient/family dissatisfaction; 2) ineffective passing of important information day to day and week to week; and 3) delayed decision-making. These latter two potential consequences may, in turn, contribute to prolonged length of stay (LOS).

For these reasons, the investigators propose a randomized control trial to test whether primary intensivists and primary nurses can decrease PICU LOS for long-stay patients. A primary intensivist is one that remains a consistent physician-presence for the patient/family and PICU team throughout the child's PICU stay, despite changes in the intensivist(s) who orchestrates day-to-day management. Primary nurses are a team of PICU nurses who provide the all/most of the bedside care to the child. The investigators hypothesize that the long-stay PICU patients who are randomized to receive primary intensivists and nurses will have a statistically lower LOS than those patients who do not.

ELIGIBILITY:
Inclusion Criteria:

* PICU patients of any age who

  * have a complex chronic condition
  * have been admitted to the PICU for one week and are predicted by the PICU attending to continue to be admitted for at least another 3 days.

Exclusion Criteria:

-

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2018-02-01 (Actual); Primary Completion 2020-02-03 (Actual); Study Completion 2020-02-03 (Actual)

PRIMARY OUTCOMES:
PICU length of stay | Up to 2 years
  Total number of days in which an individual stays in the PICU

SECONDARY OUTCOMES:
Family satisfaction | Up to 2 years
  In order to assess family satisfaction, families of all PICU patients (with PICU lengths of stay > 10 days) will be asked to complete a short anonymous questionnaire (Likert Scale) at the time of ICU discharge or within a few days when the patient is still hospitalized, if discharged late at night or over a weekend.
Provider satisfaction | Up to 2 years
  In order assess provider satisfaction, all PICU attendings, fellows, and nurses will be verbally consented and asked to complete a short anonymous questionnaire (Likert Scale) at one of two time points-1) at the end of the study or 2) before the staff member leaves
Percentage of family meetings attended by a primary nurse | Up to 2 years
  Number of meetings a nurse participated in divided by the number of meetings
Duration of invasive mechanical ventilation in those patients without chronic respiratory failure and who are on invasive mechanical ventilation from the time of enrollment | Up to 2 years
  Measured in days.
Time to tracheotomy in those who undergo a tracheotomy | Up to 2 years
  Measured in days.
Incidence of nursing-related KEEPSAFE reports recorded after enrollment | Up to 2 years
  total number of reports that are recorded.
Timing of involvement of Patient Care Services | Up to 2 years
  Measured in days.
Incidence of ICU-acquired infections after enrollment | Up to 2 years
  Total number of ICU-acquired infections
Number of documented family meetings | Up to 2 years
  Total number of family meetings.
Incidence of unplanned re-admissions to a PICU within 48 hours of PICU discharge | Up to 2 years
  Total number of unplanned re-admissions to a PICU.
Percentage of primary intensivists who meet with families | Up to 2 years
  Measured by total number of meeting divided by the number of weeks after enrollment.
Total number of shifts that are not being covered by a primary nurse, | Up to 2 years
  The Bice-Boxerman Continuity of Care Index will be used to measure continuity compliance in terms of the total number of shifts not covered by a primary nurse.

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Edwards, MD, Principal Investigator — Columbia University
Locations (1):
- Columbia University Medical Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No